CLINICAL TRIAL: NCT05596565
Title: The Effects of Observer Presence and Type on Patients' Perception of Exercise in Patients With Soft Tissue Sarcoma -A Qualitative Study
Brief Title: The Effects of Observer Presence and Type on Patients' Perception of Exercise in Patients With Soft Tissue Sarcoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Emel Mete, Research Assistant, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Qualitative study-2
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Soft Tissue Sarcoma
Keywords: soft tissue sarcoma; exercise; Telerehabilitation
MeSH Terms: conditions — Sarcoma; Motor Activity

STUDY DESIGN:
Intervention Model Description: An exploratory-descriptive qualitative study will be conducted. There will be three groups in the study with each of them will consist of ten participants. Within the scope of the study, each group will perform a similar exercise program, 2 sessions a week, for 6 weeks, in one of the 3 groups below; Group
  1. Exercising under the supervision of a face-to-face physiotherapist, Group
  2. Exercise under the observation of the physiotherapist via video-conference (telerehabilitation), Group 3: Exercising in the absence of the observer (home based exercise program).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): Supervised Exercise by a physiotherapist via face to face Participants in this group will be included in an exercise program for 6 weeks, 2 days a week and 45 minutes each session with supervised by a physiotherapist via face to face. The exercises will focus on breathing exercises, passive range of motion exercises and strengthening exercises.
  Interventions: Other: Supervised Exercise by a physiotherapist via face to face
- Experimental group 2 (Experimental): Supervised Exercise by a physiotherapist via video conference Participants in this group will be included in an exercise program for 6 weeks, 2 days a week and 45 minutes each session with supervised by a physiotherapist via video conference. The exercises will focus on breathing exercises, passive range of motion exercises and strengthening exercises.
  Interventions: Other: Supervised Exercise by a physiotherapist via face to face
- Control group (No Intervention): No Intervention: Control group: Unsupervised exercise Home based exercises will be explained to the patients and they will be asked to perform these exercises 2 days a week for 6 weeks.

INTERVENTIONS:
Other: Supervised Exercise by a physiotherapist via face to face — Participants in group-1 will be included in an exercise program for 6 weeks, 2 days a week and 45 minutes each session with supervised by a physiotherapist via face to face.
  Participants in group-2 will be included in an exercise program for 6 weeks, 2 days a week and 45 minutes each session with supervised by a physiotherapist via video conference
  Other Names: Supervised Exercise by a physiotherapist via video conference
  Arms: Experimental group 1; Experimental group 2

SUMMARY:
The primary aim of the study is to investigate the effects of supervised exercise, telerehabilitation and home-based exercise on patient perception in patients with soft tissue sarcoma. The secondary aim of the study is to identify the barriers to starting exercise in these patients.

DETAILED DESCRIPTION:
An exploratory-descriptive qualitative study will be conducted. There will be three groups in the study with each of them will consist of ten participants. Within the scope of the study, each group will perform a similar exercise program, 2 sessions a week, for 6 weeks, in one of the 3 groups below; Group 1: Exercising under the supervision of a face-to-face physiotherapist, Group 2: Exercise under the observation of the physiotherapist via video-conference (telerehabilitation), Group 3: Exercising in the absence of the observer (home based exercise program). The exercises to be applied to the groups will include breathing exercises, passive range of motion exercises and strengthening exercises. Semi-structured focus group interviews will be held with the participants twice, before and after the 6-week exercise program. In the semi-structured focus group interviews, the same questions will be asked to all participants and the verbal answers to these questions will be recorded with voice recorders. Compared to taking notes by hand; It will be preferable to record the conversation with a voice recorder because it has advantages such as recording all the interviews and allowing the interviewer to focus on the interview. In the pre-exercise interview, questions will be asked to determine the patient's views about exercises and the barriers to starting the exercise. In the interview held at the end of the exercise program, questions will be asked to learn the views/perceptions of the patients about the results of the exercise program. Thematic analysis method will be used in the evaluation of the data.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 65,
* Individuals without communication problems,
* Individuals who have been diagnosed with soft tissue sarcoma
* ECOG score ≤2

Exclusion Criteria:

* Uncontrollable arrhythmia and/or hypertension
* Presence of advanced sensory deficit
* Visual and hearing problems
* Not having sufficient communication skills (Mini Mental Test score below 24 points)
* ECOG score>2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-10 (Estimated); Primary Completion 2023-07-10 (Estimated); Study Completion 2023-09-10 (Estimated)

PRIMARY OUTCOMES:
Semi-structured focus group interviews about Patients' Perception of Exercise | Change from baseline Patients' Perception of Exercise at week 6
  Semi-structured focus group interviews will be held with the participants twice, before and after the 6-week exercise program. . In the semi-structured focus group interviews, the same questions will be asked to all participants and the verbal answers to these questions will be recorded with voice recorders. In the pre-exercise interview, questions will be asked to determine the patient's views about exercises and the barriers to starting the exercise. In the interview held at the end of the exercise program, questions will be asked to learn the views/perceptions of the patients about the results of the exercise program.

CONTACTS AND LOCATIONS:
Locations (1):
- Emel Mete, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No